CLINICAL TRIAL: NCT07038382
Title: A Randomized, Controlled, Multicenter Phase II Clinical Study to Evaluate the Efficacy, Safety, and Tolerability of HLX79 (Human Sialidase Fusion Protein) in Combination With Rituximab Injection (HLX01, Anti-CD20 Antibody) Versus Placebo in Patients With Active Glomerulonephritis
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of Human Sialidase Fusion Protein (HLX79) in Combination With Rituximab Injection Versus Placebo in Patients With Active Glomerulonephritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: HLX01HLX79-GN201
Record Dates: First submitted 2025-05-29; First posted 2025-06-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Membranous Nephropathy; Lupus Nephritis (LN)
MeSH Terms: conditions — Glomerulonephritis, Membranous; Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A1 (Experimental)
  Interventions: Drug: HLX79 10mg/kg/Placebo+HLX01
- Group B1 (Experimental)
  Interventions: Drug: HLX79 20mg/kg/Placebo + HLX01
- Group C1 (Experimental)
  Interventions: Drug: HLX79 30mg/kg/placebo+HLX01

INTERVENTIONS:
Drug: HLX79 10mg/kg/Placebo+HLX01 — Subjects with MN will receive HLX79 10mg/kg or placebo, combine with HLX01 375 mg/m2
  Arms: Group A1
Drug: HLX79 20mg/kg/Placebo + HLX01 — Subjects with MN will receive HLX79 20mg/kg or placebo combined with HLX01 375 mg/m2
  Arms: Group B1
Drug: HLX79 30mg/kg/placebo+HLX01 — Subjects with MN will receive HLX79 30mg/kg or placebo combined with HLX01 375 mg/m2
  Arms: Group C1

SUMMARY:
The primary objectives of this clinical trial is to evaluate the safety and tolerability of HLX79 in combination with HLX01 versus placebo in combination with HLX01 in the treatment of glomerulonephritis.

The secondary objective are to evaluate the pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of HLX79 and HLX01, the clinical efficacy, the dynamic changes of biomarkers of HLX79 in combination with HLX01 in the treatment of glomerulonephritis.

The subjects will receive different doses of HLX79 (10, 20, or 30 mg/kg) or placebo, all in combination with HLX01. After the end of the first treatment period, subjects will enter a 20-week follow-up period and then undergo pre-second treatment period assessments. If the investigator determines that the subject does not require the second treatment period, the subject will continue in follow-up until completing the total 48-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily participate in this clinical study, fully understand and have been informed about the study, have signed the informed consent form (ICF), and are willing to follow and able to complete all study procedures.
2. Male or female, aged 18-75 years (both inclusive) at the time of signing the ICF.
3. Diagnosed with primary membranous nephropathy (MN) within 5 year prior to screening
4. If a diagnosis of primary MN is confirmed, a renal biopsy pathological diagnosis prior to screening or a renal biopsy diagnosis obtained during screening should be available, or patients with nephrotic syndrome and a positive anti-PLA2R antibody test within 6 months prior to screening; secondary MN (secondary to infection, tumor, SLE, drugs, etc.) should be excluded; subjects should have received treatment with angiotensin-converting enzyme inhibitors (ACEIs)/angiotensin II receptor blocker (ARBs) at the highest tolerated dose judged by the investigator for 3 months prior to screening (unless intolerance to ACEI/ARB, contraindications to their use or a low blood pressure that could induce side effects, at the investigator's discretion) and also meet one of the following high-risk criteria:

   * Urine protein > 8 g/24 h at screening.(The above 3-month ACEI/ARB treatment observation period is not required)
   * eGFR ≥ 60 mL/min/1.73 m2 and urine protein > 3.5 g/24 h at screening
5. Women of childbearing potential (WOCBP) must undergo a pregnancy test at screening and obtain a negative result.
6. WOCBP or male subjects must agree to take effective contraceptive measures starting from signing the ICF until 12 months after the last dose of the investigational medicinal product (IMP).

Exclusion Criteria:

1. Pregnant or lactating women, or those with a positive blood pregnancy test prior to randomization.
2. WOCBP or partners of male subjects who plan to become pregnant during the study.
3. History of drug or alcohol abuse within 1 year prior to screening.
4. Malignancy or increased risk of malignancy prior to screening: suspected and/or diagnosed with any malignancy (except for basal cell carcinoma, squamous cell carcinoma of skin in situ, or cervical carcinoma in situ occurring within 5 years prior to screening with no evidence of recurrence after treatment).
5. History of organ transplantation or stem cell or bone marrow transplantation prior to screening, or plan to undergo the above-mentioned transplantations during the study.
6. Complicated with primary immunodeficiency diseases, type 1 diabetes mellitus, and type 2 diabetes mellitus (Type 2 diabetic patients with a renal biopsy report within one year prior to screening that excludes diabetic nephropathy are eligible to participate in this study) before screening.
7. Presence of the following diseases that are significantly unstable or poorly controlled at screening: cardiovascular disorder, hematological disease, respiratory disorder, digestive system disorder, endocrine and metabolic system disease, nervous system disorder or psychiatric disorders, skin and subcutaneous tissue disorders, musculoskeletal system disorder, immune system disorders, or Grade 3 or greater medical abnormalities (CTCAE v5.0), and the investigator believes that the subject should be excluded due to the above diseases or abnormalities, or the investigator believes that the above diseases or abnormalities may interfere with the interpretation of the study results.
8. End-stage renal disease requiring kidney transplantation or dialysis, or oliguria (urine volume < 400 mL/24 h) at screening or prior to randomization.
9. Acute, recurrent, or chronic infection (including but not limited to tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster, or atypical mycobacterial infection) at screening,
10. Infection requiring intravenous or intramuscular injection of anti-infective drugs within 2 months prior to randomization, or infection requiring hospitalization within 2 months prior to randomization.
11. Lung CT or chest X-ray at screening suggesting tuberculosis infection or previous tuberculosis infection.
12. Abnormalities in 12-lead ECG at screening, such as corrected QT (QTc) interval > 450 ms in males and corrected QT (QTc) interval > 470 ms in females (Fridericia's method).
13. Abnormal results of the following laboratory tests at screening:

    1. Hemoglobin < 90 g/L, or platelet count < 100 × 109 L, or neutrophil count < 1.5 × 109 L.
    2. Alkaline phosphatase (ALP) > 2 × upper limit of normal (ULN), or total bilirubin (TB) > 2 × ULN, or alanine aminotransferase (ALT) > 2 × ULN, or aspartate aminotransferase (AST) > 2 × ULN, or blood amylase > 1.5 × ULN.
    3. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2.
    4. International normalized ratio (INR) > 2.5 (not on anticoagulant therapy).
    5. Interferon gamma release assay positive.
    6. Serological test positive for human immunodeficiency virus (HIV) antibodies.
    7. Test results positive for treponema pallidum (syphilis).
    8. Positive for hepatitis B virus (HBV) surface antigen (HBsAg), or positive for HBV core antibody (HBcAb) and HBV deoxyribonucleic acid (HBV-DNA).
    9. Hepatitis C virus (HCV) infection (HCV antibody positive with HCV-RNA > ULN).
14. History of serious drug allergy before screening: history of allergy to two or more drugs, or history of allergy or serious side effects to HLX01, HLX79, or their excipients, or history of anaphylaxis to intravascular injection of contrast agents, human or murine proteins, or monoclonal antibodies, or history of anaphylactic shock.
15. History of or need for treatment with one of the following drugs prior to screening:

    * Treatment with glucocorticoids, MMF (or other forms of mycophenolate) within 1 month prior to randomization
    * Treatment with calcineurin inhibitors (CNIs) such as tacrolimus and cyclosporine A or other immunosuppressive agents within 3 months prior to randomization
    * Treatment with alkylating agents such as cyclophosphamide (CYC) and ifosfamide within 6 months prior to randomization
    * Subjects who still require treatment with glucocorticoids, MMF (or other forms of mycophenolate), or alkylating agents or other immunosuppressive agents during the study as judged by the investigator at screening.
16. Have received treatment with abatacept, telitacicept, JAK inhibitors, thalidomide, lenalidomide, bortezomib, cladribine, belimumab, rituximab, or other targeted drugs (T lymphocytes, B lymphocytes, interleukin-1, interleukin-6, type I interferon, etc.) within 1 year prior to randomization.Subjects who have received B-cell depleting drugs (such as rituximab) within the past year are eligible to participate in this study if there is evidence that the number of CD19+ or CD20+ B cells have recovered to the lower limit of normal or above.
17. Have received intravenous infusion of immunoglobulin or plasma exchange within 3 months prior to randomization.
18. Have participated in a clinical study of other investigational medicinal products prior to screening, with an interval between this study and the previous study being too short: within 1 month prior to the first administration of this study or within 5 half-lives of the previous investigational medicinal product (whichever is longer). Or plan to participate in clinical studies of other investigational medicinal products before completing all scheduled assessments in this clinical study.
19. Have participated in surgical or device clinical studies within 3 months prior to screening or plan to participate in other surgical or device clinical studies during this clinical study.
20. Have received any live or live attenuated vaccine within 3 months prior to screening, or plan to receive any live or live attenuated vaccine during the study.
21. Use of herbal medicines, traditional Chinese medicines, or local traditional remedies that have therapeutic effects for MN within 14 days prior to randomization.
22. Unable to establish venous access due to poor tolerability or difficulty in finding veins, or unable or unwilling to undergo repeated venipuncture.
23. Donated whole blood or blood components (more than 400 mL) or lost a large amount of blood (more than 400 mL) within 2 months prior to screening, or plan to donate whole blood or blood components during the study.
24. The investigator has a clear reason to believe that participation in this study will damage the rights and interests of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 24 weeks
  Including incidence, nature, and severity of adverse events (AEs) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0, and the incidence of serious adverse events (SAEs), adverse events of special interest (AESIs), abnormal laboratory tests, vital signs, physical examination, and 12-lead ECG

SECONDARY OUTCOMES:
Assessment of safety | 52 weeks
  Safety: Proportion of subjects with at least one Grade 3 or greater infection-related AE in each dose group according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE, and higher grades mean a worse outcome.
Plasma concentrations and PK parameters of HLX79 and HLX01 | 52 weeks
  Peak concentration (Cmax, Cmax, ss)
Plasma concentrations and PK parameters of HLX79 and HLX01 | 52 weeks
  Time to peak (Tmax, Tmax, ss)
Plasma concentrations and PK parameters of HLX79 and HLX01 | 52 weeks
  Area under the concentration-time curve (AUC0-inf, AUC0-t, AUC0-tau, AUCss)
Plasma concentrations and PK parameters of HLX79 and HLX01 | 52 weeks
  Elimination half-life (t1/2, t1/2, ss)
Plasma concentrations and PK parameters of HLX79 and HLX01 | 52 weeks
  Clearance (CL, CLss)
Plasma concentrations and PK parameters of HLX79 and HLX01 | 52 weeks
  Volume of distribution (Vz, Vss)
Plasma concentrations and PK parameters of HLX79 and HLX01 | 52 weeks
  Accumulation ratio (Rac)
PD | 52 weeks
  Proportion of subjects with peripheral blood CD19+ B lymphocyte count ≤ 5/μL at weeks 12, 24, 36, and 52 of treatment, and proportion of subjects with peripheral blood CD20+ B lymphocyte count ≤ 1/μL at weeks 12, 24, 36, and 52 of treatment
Immunogenicity evaluation | 52 weeks
  Positive rates of anti-drug antibody (ADA) and neutralizing antibody (NAb, if applicable) for HLX79 and HLX01
Assessment of clinical efficacy | 52 weeks
  Proportion of subjects achieving complete remission (CR) or partial remission (PR) at weeks 12, 24, 36, and 52 of treatment.
Assessment of clinical efficacy | 52 weeks
  Proportion of subjects negative for anti-M-type phospholipase A2 receptor (PLA2R) antibodies at weeks 12, 24, 36, and 52 of treatment.
Assessment of clinical efficacy | 52 weeks
  Changes in anti-PLA2R antibody level from baseline at weeks 12, 24, 36, and 52 of treatment.
Explore the biomarkers | 52 weeks
  Peripheral blood B lymphocyte counts or B lymphocyte kinetics: including the depletion kinetics of B lymphocytes and their subsets (CD20+ B lymphocytes, CD19+ B lymphocytes, and memory B lymphocytes)
Explore the biomarkers | 52 weeks
  Peripheral blood B lymphocyte counts or B lymphocyte kinetics: the recovery kinetics of B lymphocytes and their subsets (e.g., CD20+ B lymphocytes, CD19+ B lymphocytes, and memory B lymphocytes).
Explore the biomarkers | 52 weeks
  Serum immunoglobulins (IgA, IgG, and IgM).
Explore the biomarkers | 52 weeks
  Serum complements (C3 and C4).
Explore the biomarkers | 52 weeks
  Urine CD163

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Beijing Tsinghua Changgung Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Xiangya Hospital Of Gentral South University, Changsha
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital Zhejiang University School Of Medicine, Hangzhou
  - The Second Hospital of Anhui Medical University, Hefei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Jiangxi Provincial People's Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Zhongdong Hospital Southeast University, Nanjing
  - Shanghai General Hospital, Shanghai
  - Renmin Hospital Of Wuhan University, Wuhan
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an
  - The First Affiliated Hospital Of Xiamen University, Xiamen
  - Su Bei People's Hospital, Yangzhou

IPD SHARING:
Plan to Share IPD: No